CLINICAL TRIAL: NCT01327638
Title: Safety Data on Etoricoxib From Swedish Registries of Spondyloarthropathy/Ankylosing Spondylitis Patients
Brief Title: Safety of Etoricoxib (MK-0663) in Patients With Spondyloarthropathy (SpA)/Ankylosing Spondylitis (AS) in Sweden (EP07013.013.11.082)
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: 0663-159; EP07013.013.11.082 (Other: Merck)
Record Dates: First submitted 2011-03-11; First posted 2011-04-01 (Estimated); Last update posted 2024-05-10 (Actual); Status verified 2022-02

CONDITIONS: Spondylarthropathies; Spondylitis, Ankylosing
MeSH Terms: conditions — Spondylarthropathies; Spondylitis | interventions — Etoricoxib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients with SpA/AS and etoricoxib treatment
  Interventions: Drug: etoricoxib
- Patients with SpA/AS and other COX-2 inhibitor treatment
  Interventions: Drug: Other COX-2 inhibitor
- Patients with SpA/AS and nsNSAIDs treatment
  Interventions: Drug: nsNSAIDs

INTERVENTIONS:
Drug: etoricoxib — Patients with SpA/AS who took etoricoxib
  Other Names: MK-0663; Arcoxia
  Groups: Patients with SpA/AS and etoricoxib treatment
Drug: Other COX-2 inhibitor — Patients with SpA/AS who took other COX-2 inhibitors
  Groups: Patients with SpA/AS and other COX-2 inhibitor treatment
Drug: nsNSAIDs — Patients with SpA/AS who took nsNSAIDs
  Groups: Patients with SpA/AS and nsNSAIDs treatment

SUMMARY:
The study is intended to provide additional post-marketing safety data regarding the use of etoricoxib for the indication of ankylosing spondylitis.

DETAILED DESCRIPTION:
The specific project objectives are to:

1) Describe the characteristics of Swedish patients with inflammatory SpA/AS ; 2) Describe the use of etoricoxib and other cyclooxygenase-2 (COX-2 inhibitors)/non-selective nonsteroidal anti-inflammatory drugs (nsNSAIDs) in Swedish patients with SpA/AS; and 3) Estimate and compare the rates of clinical outcomes of special interest (gastrointestinal, renovascular, cardiovascular and cerebrovascular) with use of etoricoxib and other COX-2 inhibitors/nsNSAIDs in Swedish patients with SpA/AS. Comparisons of clinical outcomes among the drugs of interest will be made by descriptive comparison of the point estimates for the incidence rates and their associated 95% confidence intervals (CIs), using both clinical and epidemiological judgment and in light of the limitations of this observational study. No formal statistical significance testing will be performed for purposes of such comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Participant attended an out-patient clinic 2001-2010.
* Participant is registered with an International Classification of diseases (ICD, Version 10)-code corresponding to SpA/AS and AS.

Exclusion Criteria:

Not applicable.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Out-patients in Sweden with SpA/AS who took etoricoxib, other COX-2 inhibitors, or nsNSAIDs from 2001-2010.
Sampling Method: Probability Sample
Enrollment: 21108 (Actual)
Dates: Start 2011-02-15 (Actual); Primary Completion 2018-09-24 (Actual); Study Completion 2018-12-06 (Actual)

PRIMARY OUTCOMES:
Number of patients with Characteristics of inflammatory SPA/AS | Over a 12 year period (2001-2013)
Number of patients who used etoricoxib | Up to 7 1/2 years (Q3 2005 - 2013)
Number of patients who used other COX-2 inhibitors | Up to 7 1/2 years (Q3 2005 - 2013)
Number of patients who used nsNSAIDs | Up to 7 1/2 years (Q3 2005 - 2013)
Number of clinical outcomes of special interest | Up to 7 1/2 years (Q3 2005 - 2013)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: EU PAS Register (EUPAS19202) — http://www.encepp.eu/encepp/viewResource.htm?id=27099